CLINICAL TRIAL: NCT05964894
Title: Occupational Therapy for Work-related Musculoskeletal Disorders Among Hemodialysis Nurse
Brief Title: An Ergonomic Training With Exercise Program for Work-related Musculoskeletal Disorders Among Hemodialysis Nurse
Acronym: WMSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jer-Hao Chang (Other)
Responsible Party: Sponsor-Investigator, Jer-Hao Chang, Associate Professor, National Cheng-Kung University Hospital
Organization: National Cheng-Kung University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: A-ER-108-235
Record Dates: First submitted 2023-07-10; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Musculoskeletal Disorders
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ergonomic training group (Experimental): The ergonomic training group received a 12-week ergonomic training program.
  Interventions: Other: ergonomic training
- No training group (No Intervention): The no training group did not receive any training program.

INTERVENTIONS:
Other: ergonomic training — ergonomic education & exercise training
  Arms: Ergonomic training group

SUMMARY:
This study aimed to examine the effectiveness of the 12-week ergonomic intervention developed by Person-Environment-Occupation (PEO) model in improving musculoskeletal discomfort and muscle strength for hemodialysis nurses. The maintenance effects of the intervention were also evaluated after another 12-week follow-up.

DETAILED DESCRIPTION:
Methods A cluster experimental design was used to conduct this study. Participants were recruited from hemodialysis units at two medical centers in Taiwan and had complaints of work-related musculoskeletal disorders (WMSDs) within the past six months. By PEO model, the 12-week intervention including ergonomic education and exercise program was designed based on the job contents of hemodialysis nurses. In the study period, we used a mobile massager app to reminder them and monitor their implementation of exercises. The outcome indicators were measured before and after intervention as well as the follow-up after another 12 weeks. A generalized estimating equations model was adopted to analyze the repeated measurements.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 65 years old, which is the legal age range of adult for work in Taiwan
* registered nurses to work full time in the hemodialysis unit more than 6 months,
* having complaint of WMSDs within previous 6 months before this study.

Exclusion Criteria:

* having no musculoskeletal disorder related to the job
* to care less than 4 patients in 4 hours, which was below the Taiwan workload reference for nurse in hemodialysis job
* to have any other consideration to keep from 12- week physical exercise program (such as pregnancy, injury, disease, leave…, etc.).

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
severity degree of muscular discomfort | week 0
  self reported by Nordic Musculoskeletal Questionnaire (0-5 points; the higher score indicates the more discomfort)
muscle strength | week 0
  grip and pinch power; the muscle strength of neck extension, shoulder flexion/extension, and wrist flexion/extension of the dominant (maximal force of the muscles movement against in kilograms, the higher the stronger)
severity degree of muscular discomfort | week 12
  self reported by Nordic Musculoskeletal Questionnaire (0-5 points; the higher score indicates the more discomfort)
muscle strength | week 12
  grip and pinch power; the muscle strength of neck extension, shoulder flexion/extension, and wrist flexion/extension of the dominant (maximal force of the muscles movement against in kilograms, the higher the stronger)
severity degree of muscular discomfort | week 24
  self reported by Nordic Musculoskeletal Questionnaire (0-5 points; the higher score indicates the more discomfort)
muscle strength | week 24
  grip and pinch power; the muscle strength of neck extension, shoulder flexion/extension, and wrist flexion/extension of the dominant (maximal force of the muscles movement against in kilogram, the higher the stronger)

SECONDARY OUTCOMES:
Subjective quality of life | week 0
  World Health Organization Quality of Life, Brief edition, Taiwan version (1-5, higher score for higher quality of life)
Subjective quality of life | week 24
  World Health Organization Quality of Life, Brief edition, Taiwan version (1-5, higher score for higher quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: JER-HAO CHANG, PH.D., Principal Investigator — National Cheng Kung University, College of Medicine
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No